CLINICAL TRIAL: NCT06009146
Title: Results of Endovascular Treatment for Infrapopliteal Arterial Occlusive Disease: a Prospective, Multicenter, Real-world Study
Brief Title: Results of Endovascular Treatment for Infrapopliteal Arterial Occlusive Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Peking University Third Hospital (Other); Peking University First Hospital (Other); Beijing Hospital (Other Government); Chengdu University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Dalian Medical University (Other); Huashan Hospital (Other); Shanghai Pudong Hospital (Other); Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Changhai Hospital (Other); Hebei General Hospital (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); LanZhou University (Other); The Second Hospital University of South China (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Affiliated Hospital of Qingdao University (Other); Qingdao Haici Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other); First Hospital of Tsinghua University (Other); Shanxi Provincial People's Hospital (Other Government); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); RenJi Hospital (Other); The Luhe Teaching Hospital of the Capital Medical University (Other); Beijing Friendship Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Tianjin First Central Hospital (Other); Tianjin Medical University General Hospital (Other); Renmin Hospital of Wuhan University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Zhejiang University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IPOD-Real Study
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Infrapopliteal Artery Occlusive Disease; Endovascular Treatment
Keywords: Endovascular Treatment; Infrapopliteal Artery Disease; Drug-coated Balloons; Angioplasty; Atherectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rutherford scale < 4
  Interventions: Device: Endovascular treatment
- Rutherford scale 4-5
  Interventions: Device: Endovascular treatment
- Rutherford scale 6
  Interventions: Device: Endovascular treatment

INTERVENTIONS:
Device: Endovascular treatment — Endovascular treatment for infrapopliteal arterial disease.

SUMMARY:
This study is a prospective, multi-center observational study, which evaluates the effectiveness and safety of endovascular therapy in the real world for infrapopliteal arterial occlusive disease from intermittent claudication to chronic threatening limb ischemia.

DETAILED DESCRIPTION:
This study is a prospective, multi-center observational study. This study will be conducted at 38 centers and is expected to enroll more than 3000 patients. And we will evaluate the effectiveness and safety of endovascular therapy in the real world for infrapopliteal arterial occlusive disease from intermittent claudication to chronic threatening limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥ 18 years of age; Patients with ≥1 infrapopliteal artery disease (P3 popliteal artery, anterior tibial artery, posterior tibial artery, peroneal artery, tibiofibular trunk) need to receive endovascular treatment, regardless of whether there is a combination of supra-knee or submalleolar occlusion; Patients voluntary and capable of follow-up;

Exclusion Criteria:

Patients who are known to be allergic to heparin, aspirin, other antiplatelet drugs, contrast agents, etc., and those who are unable to undergo endovascular therapy for other reasons; Pregnant and lactating women; Patients with thromboangiitis obliterans；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infrapopliteal arterial occlusive disease undergoing endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from major adverse event rate | 12 months
  Major adverse events include Death, major amputation rates and clinical driven target lesion revascularization (CDTLR).

SECONDARY OUTCOMES:
Amputation-free survival | 12 months
  Freedom from death and major amputation
Survival | 12 months
  Freedom from all-cause mortality.
Freedom from major amputation | 12 months
  Freedom from major amputation
Freedom from CDTLR | 12 months
  Freedom from clinical driven target lesion revascularization
Freedom from clinical driven target limb revascularization | 12 months
  Freedom from clinical driven target limb revascularization
Rutherford categories | 12 months
  Rutherford categories
Wound condition | 12 months
  Wound and foot infections were scored using WIfI system.
Complication rates | 1 week
  Minor and Major complications rates.
Quality of life score | 12 months
  Vascular quality of life questionnaire was used.

CONTACTS AND LOCATIONS:
Overall Officials: Lianrui Guo, M.D., Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided